CLINICAL TRIAL: NCT05171777
Title: A Randomized, Multicenter, Open-Label Cross-Over Study to Evaluate Participant and Healthcare Professional Reported Preference for Subcutaneous Atezolizumab Compared With Intravenous Atezolizumab Formulation in Participants With Non-Small Cell Lung Cancer
Brief Title: A Study to Evaluate Participant and Healthcare Professional Reported Preference for Subcutaneous Atezolizumab Compared With Intravenous Atezolizumab Formulation in Participants With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MO43576
Record Dates: First submitted 2021-11-29; First posted 2021-12-29 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Participants will receive atezolizumab SC followed by atezolizumab IV.
  Interventions: Drug: Atezolizumab
- Treatment B (Experimental): Participants will receive atezolizumab IV followed by atezolizumab SC.
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered on Day 1 of each 21-day cycle. Participants will receive atezolizumab according to their assigned route of administration (i.e., SC or IV) for the first three treatment cycles. At Cycle 4, participants will cross-over and receive atezolizumab administered according to the alternative route of administration for Cycles 4-6. This period of 3+3 cycles in both treatment arms constitutes the study Treatment Cross-over Period. After Cycle 6, participants will select how they would like atezolizumab to be administered (SC or IV) for the Treatment Continuation Period. The Treatment Continuation Period will continue until Cycle 16 for participants with early-stage NSCLC or until loss of clinical benefit, as determined by the investigator according to local standard of care, for patients with advanced NSCLC.
  Other Names: Tecentriq

SUMMARY:
This is a Phase II, randomized, multi-center, multinational, open-label, cross-over study in adult participants with PD-L1-positive NSCLC. Two populations will be included: participants with resected Stage II, IIIA, and selected IIIB (T3-N2) NSCLC who have completed adjuvant platinum-based chemotherapy without evidence of disease relapse/recurrence, and chemotherapy-naïve participants with Stage IV NSCLC. The study will evaluate participant- and healthcare professionals (HCP)-reported preference for atezolizumab subcutaneous (SC) compared with atezolizumab intravenous (IV).

ELIGIBILITY:
Inclusion Criteria for All Participants:

* ECOG performance status of 0 or 1

Inclusion Criteria for Participants with Early-stage NSCLC:

* Participants must have a complete resection of a histologically or cytologically confirmed Stage II, IIIA, and selected IIIB (T3-N2) NSCLC
* PD-L1 expression TC ≥ 1% or TPS ≥ 1%
* Participants must have completed adjuvant chemotherapy at least 4 weeks and up to 12 weeks prior to randomization and must be adequately recovered from chemotherapy. For participants in the adjuvant setting, neoadjuvant chemotherapy or chemoradiotherapy is acceptable provided that participants also received adjuvant chemotherapy as per protocol's requirement.

Inclusion Criteria for Participants with Stage IV NSCLC:

* Histologically or cytologically confirmed, Stage IV non-squamous or squamous NSCLC
* Life expectancy ≥ 18 weeks in the opinion of the investigator
* PD-L1 expression TC ≥ 50% or TPS ≥ 50% or TC3 or IC3
* No prior systemic treatment for Stage IV non-squamous or squamous NSCLC
* Participants who have received prior neo-adjuvant, adjuvant chemotherapy, radiotherapy, or chemoradiotherapy with curative intent for non-metastatic disease must have experienced a treatment-free interval of at least 6 months from randomization since the last chemotherapy, radiotherapy, or chemoradiotherapy cycle.

Exclusion Criteria for All Participants:

* History of malignancy within 5 years prior to initiation of study treatment, with the exception of the cancer under investigation in this study and malignancies with a negligible risk of metastasis or death
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Participants known to have a sensitizing mutation in the EGFR gene or an ALK fusion oncogene
* History of leptomeningeal disease
* Uncontrolled or symptomatic hypercalcemia
* Active or history of autoimmune disease or immune deficiency
* History of idiopathic pulmonary fibrosis, organizing pneumonia), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Significant cardiovascular disease within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina

Exclusion Criteria for Participants with Stage IV NSCLC:

* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (36):
- United States (4):
  - New Jersey Hematology Oncology Associates LLC, Brick, New Jersey
  - Tri County Hematologyoncology, Massillon, Ohio
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - UPMC - Hillman Cancer Center, Pittsburgh, Pennsylvania
- Argentina (3):
  - Fundación CENIT para la Investigación en Neurociencias, Buenos Aires
  - CEMIC, Buenos Aires
  - Centro Oncologico Korben, Ciudad Autonoma Buenos Aires
- Brazil (4):
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
- Canada (2):
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - Sault Area Hospital, Sault Ste. Marie, Ontario
- OrlandiOncología, Santiago, Chile
- Costa Rica (2):
  - Clinica CIMCA, San José
  - ICIMED Instituto de Investigación en Ciencias Médicas, San José
- Finland (4):
  - Oulun yliopistollinen sairaala (OYS), Oulu
  - Tampereen yliopistollinen sairaala (TAYS), Tampere
  - Turun yliopistollinen keskussairaala (TYKS), Turku
  - Vaasan Keskussairaala, Vaasa
- Italy (4):
  - Azienda Ospedaliera Universitaria Senese, Siena, Abruzzo
  - IRCCS Istituto Regina Elena (IFO), Rome, Lazio
  - Instituto Europeo di Oncologia, Milan, Lombardy
  - A.O.U. Maggiore della Carità, Novara, Piedmont
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, R?ga
  - Riga East Clinical University Hospital Latvian Oncology Centre, Riga
- Poland (2):
  - Warminsko-Mazurskie Centrum Chorób P?uc w Olsztynie, Olsztyn
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy, Otwock
- South Korea (2):
  - Chungbuk National University Hospital, Cheongju-si
  - Asan Medical Center, Seoul
- Spain (6):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña, LA Coruna
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Majem M, Chewaskulyong B, Zvirbule Z, Lee KH, Korbenfeld E, Kolb-Sielecki J, Castro Sanchez AY, Bustillos A, Herraez-Baranda L, Liu X, Kim SW, Cappuzzo F. Exploratory Analyses of Patient Preferences for Atezolizumab Subcutaneous Versus Intravenous from the IMscin002 Study in Patients with Non-Small Cell Lung Cancer. Oncol Ther. 2025 Nov 26. doi: 10.1007/s40487-025-00402-x. Online ahead of print. PMID 41296193

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study across 37 investigative sites in 12 countries (Spain, Brazil, Finland, Italy, United States, Argentina, Canada, Republic of Korea, Costa Rica, Latvia, Poland, and Chile) from 04 April 2022 to 25 October 2024.
Pre-assignment Details: A total of 179 participants with non-small cell lung cancer (NSCLC) were randomized in 1:1 ratio to Arm A (atezolizumab IV followed by atezolizumab SC) or Arm B (atezolizumab SC followed by atezolizumab IV). The study consists of two periods: Treatment Crossover Period, and Treatment Continuation Period.
Groups:
- Crossover Atezolizumab IV/SC: Participants were administered atezolizumab, intravenous (IV) infusion, 1200 milligrams (mg), every 3 weeks (Q3W) for 3 cycles followed by atezolizumab, subcutaneous (SC) injections, 1875 mg, Q3W, for the next 3 cycles (cycle length=21 days) in the Treatment Crossover Period.
- Crossover Atezolizumab SC/IV: Participants were administered atezolizumab, SC injections, 1875 mg, Q3W for 3 cycles followed by atezolizumab, IV, 1200 mg, Q3W, for the next 3 cycles (cycle length=21 days) in the Treatment Crossover Period.
- Continuation Atezolizumab IV: After 6 cycles of treatment in Crossover Period, participants were given an option to choose between IV or SC administration of atezolizumab for the Treatment Continuation Period. Participants in this arm chose to continue treatment with atezolizumab IV, 1200 mg Q3W up to Cycle 16 for participants with early-stage NSCLC or until loss of clinical benefit for participants with advanced NSCLC.
- Continuation Atezolizumab SC: After 6 cycles of treatment in Crossover Period, participants were given an option to choose between IV or SC administration of atezolizumab for the Treatment Continuation Period. Participants in this arm chose to continue treatment with atezolizumab SC, 1875 mg Q3W up to Cycle 16 for participants with early-stage NSCLC or until loss of clinical benefit for participants with advanced NSCLC.
Period: Treatment Crossover Period
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Started | 89 | 90 | 0 | 0
Completed | 55 | 60 | 0 | 0
Not Completed | 34 | 30 | 0 | 0
Not completed — Adverse Event | 9 | 6 | 0 | 0
Not completed — Death | 5 | 5 | 0 | 0
Not completed — Disease Relapse | 1 | 0 | 0 | 0
Not completed — Reason not Specified | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 14 | 10 | 0 | 0
Not completed — Protocol Violation | 0 | 2 | 0 | 0
Not completed — Symptomatic Deterioration | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 0 | 0
Period: Treatment Continuation Period
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Started | 0 | 0 | 26 | 89
Completed | 0 | 0 | 11 | 32
Not Completed | 0 | 0 | 15 | 57
Not completed — Adverse Event | 0 | 0 | 3 | 6
Not completed — Death | 0 | 0 | 1 | 3
Not completed — Disease Relapse | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 4
Not completed — Progressive Disease | 0 | 0 | 6 | 20
Not completed — Study Ended by Sponsor | 0 | 0 | 4 | 15
Not completed — Symptomatic Deterioration | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 6

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants.
Groups:
- Crossover Atezolizumab IV/SC: Participants were administered atezolizumab, IV infusion, 1200 mg, Q3W for 3 cycles followed by atezolizumab, SC injections, 1875 mg, Q3W, for the next 3 cycles (cycle length=21 days) in the Treatment Crossover Period.
- Total: Total of all reporting groups
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Total
Number analyzed (Participants) | 89 | 90 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (9.2) | 67.7 (9.4) | 67.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 32 | 60
  Male | 61 | 58 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 18 | 38
  Not Hispanic or Latino | 55 | 62 | 117
  Unknown or Not Reported | 14 | 10 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 5 | 8 | 13
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 75 | 74 | 149
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Preferred Atezolizumab SC to Atezolizumab IV Assessed Using Patient Preference Questionnaire (PPQ)
Description: Participants preference was assessed based on the Question 1 of PPQ. Question 1 (All things considered, which route of administration did you prefer?) asks participants to report their preference for the route of administration (IV, SC, or no preference). A point estimate with associated 95% CI for the percentage of participants who preferred atezolizumab SC was calculated. Participants experiencing any of the following events: treatment withdrawal prior to eligibility for PPQ, or death without answering Question 1 of PPQ, or treatment not started; were excluded from the analysis set. Participants who answered Question 1 of the PPQ without having at least 2 consecutive administrations of treatment with each administration modality (SC and IV) were excluded from the analysis. Percentages have been rounded off. As planned, participant preference was summarized and presented by overall (all participants) and by randomized treatment sequence using FAS.
Time Frame: Cycle 6 Day 1 (cycle length=21 days)
Population: FAS included all randomized participants. Overall number analyzed is the number of participants who answered Question 1 of PPQ.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- All Participants: Participants either received atezolizumab IV, 1200 mg for the first 3 cycles, followed by SC, 1875 mg for the next three cycles, or atezolizumab SC 1875 mg, for the first 3 cycles, followed by IV 1200 mg for the next three cycles during the Treatment Crossover Period.
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | All Participants
Number analyzed (Participants) | 60 | 63 | 123
percentage of participants | 71.67 [58.56 to 82.55] | 69.84 [56.98 to 80.77] | 70.73 [61.85 to 78.59]

2. Secondary Outcome: Number of Participants by Their Level of Satisfaction With Atezolizumab SC and Atezolizumab IV Assessed Using Therapy Administration Satisfaction Questionnaire - Subcutaneous (TASQ-SC) and Intravenous (TASQ-IV)
Description: TASQ is a 12-item, participant-reported questionnaire measuring the impact of each mode of treatment administration (TASQ-IV for IV treatment and TASQ-SC for SC treatment) on five domains: Physical Impact, Psychological Impact, Impact on Activities of Daily Living, Convenience, and Satisfaction. TASQ-IV/-SC was administered at treatment Cycles 3 and 6 according to the order of treatment received per arm during the Crossover Period. Participants satisfaction was assessed based on the Question 1 of TASQ-IV/SC which asks participants about their satisfaction with respect to route of administration (very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied, participant did not answer the question). Question 1 - TASQ- IV (How satisfied or dissatisfied were you with the IV infusion?) and TASQ- SC (How satisfied or dissatisfied were you with the SC injection?)
Time Frame: Cycles 3 Day 1 and Cycle 6 Day 1 (cycle length=21 days)
Population: FAS included all randomized participants. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants who answered Question 1 of TASQ IV/SC.
Measure: Count of Participants; unit: Participants
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV
Number analyzed (Participants) | 74 | 71
Participants
  TASQ- IV- Very Satisfied: number analyzed (Participants) | 74 | 59
  TASQ- IV- Very Satisfied | 25 | 10
  TASQ- IV- Satisfied: number analyzed (Participants) | 74 | 59
  TASQ- IV- Satisfied | 31 | 34
  TASQ- IV- Neither Satisfied nor Dissatisfied: number analyzed (Participants) | 74 | 59
  TASQ- IV- Neither Satisfied nor Dissatisfied | 17 | 11
  TASQ- IV- Dissatisfied: number analyzed (Participants) | 74 | 59
  TASQ- IV- Dissatisfied | 1 | 1
  TASQ- IV- Very Dissatisfied: number analyzed (Participants) | 74 | 59
  TASQ- IV- Very Dissatisfied | 0 | 3
  TASQ- IV- Participant did not Answer Question: number analyzed (Participants) | 74 | 59
  TASQ- IV- Participant did not Answer Question | 0 | 0
  TASQ- SC- Very Satisfied: number analyzed (Participants) | 56 | 71
  TASQ- SC- Very Satisfied | 22 | 30
  TASQ- SC- Satisfied: number analyzed (Participants) | 56 | 71
  TASQ- SC- Satisfied | 21 | 36
  TASQ- SC- Neither Satisfied nor Dissatisfied: number analyzed (Participants) | 56 | 71
  TASQ- SC- Neither Satisfied nor Dissatisfied | 9 | 5
  TASQ- SC- Dissatisfied: number analyzed (Participants) | 56 | 71
  TASQ- SC- Dissatisfied | 3 | 0
  TASQ- SC- Very Dissatisfied: number analyzed (Participants) | 56 | 71
  TASQ- SC- Very Dissatisfied | 1 | 0
  TASQ- SC- Participant did not Answer Question: number analyzed (Participants) | 56 | 71
  TASQ- SC- Participant did not Answer Question | 0 | 0

3. Secondary Outcome: Percentage of Participants Who Select Atezolizumab SC for Treatment Continuation Period
Description: At Cycle 6, Day 1, participants were expected to select the route of study treatment administration (SC or IV) they would like to receive during the Treatment Continuation Period (starting at Cycle 7). Percentage of participants who chose SC administration have been reported here. Percentages have been rounded off.
Time Frame: Cycle 6 Day 1 (Cycle length=21 days)
Population: FAS included all randomized participants. Overall number analyzed is the number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV
Number analyzed (Participants) | 55 | 60
percentage of participants | 78.2 | 76.7

4. Secondary Outcome: Duration of Treatment Preparation According to Healthcare Professionals (HCPs) Response to Perception of Time, Assessed Using Question 1 of Healthcare Professional Questionnaires (HCPQs) - Drug Preparation Area
Description: The HCPQ- Drug Preparation Area Question 1 was completed by the HCPs within the pharmacy/drug preparation area where atezolizumab IV reconstitution or atezolizumab SC was prepared before the actual drug administration took place. The HCPQs were completed for every participant at each treatment cycle (Cycles 1-6, i.e., 3 cycles of atezolizumab IV followed by 3 cycles of atezolizumab SC or vice versa) of the treatment cross-over period. HCPs responded to the following parts of Question 1 that sought to evaluate the amount of time it took to prepare the IV infusion/SC injection of atezolizumab: "How long (in minutes) did it take to prepare the treatment for use?"
Time Frame: Day 1 of Cycles 1 to 6 (cycle length= 21 days)
Population: Overall number analyzed included HCPs who completed Question 1 of the survey. The number analyzed included HCPs who completed Question 1 of the survey at the specified treatment cycles.
Measure: Median (Full Range); unit: minutes
Groups:
- Atezolizumab IV/SC: Participants were administered atezolizumab, IV infusion, 1200 mg, Q3W for 3 cycles followed by atezolizumab, SC injections, 1875 mg, Q3W, for the next 3 cycles (cycle length=21 days) in the Treatment Crossover Period. HCPs who prepared and/or administered the IV/SC formulations completed the HCPQ questionnaire
- Atezolizumab SC/IV: Participants were administered atezolizumab, SC injections, 1875 mg, Q3W for 3 cycles followed by atezolizumab, IV, 1200 mg, Q3W, for the next 3 cycles (cycle length=21 days) in the Treatment Crossover Period. HCPs who prepared and/or administered the IV/SC formulations completed the HCPQ questionnaire.
Arm/Group | Atezolizumab IV/SC | Atezolizumab SC/IV
Number analyzed (Participants) | 84 | 83
minutes
  Cycle 1 | 5.0 [1 to 40] | 5.0 [1 to 45]
  Cycle 2: number analyzed (Participants) | 80 | 80
  Cycle 2 | 5.0 [1 to 40] | 5.0 [1 to 35]
  Cycle 3: number analyzed (Participants) | 72 | 74
  Cycle 3 | 5.0 [1 to 45] | 4.5 [1 to 40]
  Cycle 4: number analyzed (Participants) | 67 | 71
  Cycle 4 | 5.0 [1 to 35] | 5.0 [1 to 50]
  Cycle 5: number analyzed (Participants) | 62 | 64
  Cycle 5 | 5.0 [1 to 35] | 5.0 [1 to 59]
  Cycle 6: number analyzed (Participants) | 56 | 60
  Cycle 6 | 5.0 [1 to 35] | 5.0 [1 to 36]

5. Secondary Outcome: Percentage of HCPs by Their Response to Perception of Impact on Clinical Management and Clinical Efficiency of Atezolizumab SC and IV, Assessed Using Question 2 of HCPQ - Drug Preparation Area
Description: HCPs within pharmacy/drug preparation area responded to HCPQ-Drug Preparation Area Question 2 at Cycle 6 of Treatment Crossover Period for every participant: "If all IV infusions are switched to SC, please indicate how strongly you agree/disagree with each of following statements: a=Staff will have increased availability for other tasks in pharmacy; b=Administrative procedures around atezolizumab SC will require less time; c=Atezolizumab SC formulations will provide more flexibility for staff in managing their workload; d=Due to ready-to-use atezolizumab SC formulations, potential dosing errors will be avoided; e=Due to ready-to-use atezolizumab SC formulations, there will be less drug wastage; f=Without having to reconstitute the drug, less storage space for atezolizumab SC related supplies will be required in pharmacy; g=Preparation procedures & associated time staff time commitment will be reduced, h=It will ease drug administration for participants with difficult venous access."
Time Frame: Cycle 6 Day 1 (cycle length=21 days)
Population: Overall number analyzed included HCPs who completed Question 2 of the survey at treatment Cycle 6. Percentages have been rounded off.
Measure: Number; unit: percentage of HCPs
Groups:
- Atezolizumab IV/ SC: Participants were administered atezolizumab, IV infusion, 1200 mg, Q3W for 3 cycles followed by atezolizumab, SC injections, 1875 mg, Q3W, for the next 3 cycles (cycle length=21 days) in the Treatment Crossover Period. HCPs who prepared and/or administered the IV/SC formulations completed the HCPQ questionnaire.
- Atezolizumab SC/ IV: Participants were administered atezolizumab, SC injections, 1875 mg, Q3W for 3 cycles followed by atezolizumab, IV, 1200 mg, Q3W, for the next 3 cycles (cycle length=21 days) in the Treatment Crossover Period. HCPs who prepared and/or administered the IV/SC formulations completed the HCPQ questionnaire.
Arm/Group | Atezolizumab IV/ SC | Atezolizumab SC/ IV
Number analyzed (Participants) | 57 | 60
percentage of HCPs
  a=Strongly Disagree | 7.0 | 10.0
  a=Disagree | 7.0 | 0
  a=Neutral | 21.1 | 31.7
  a=Agree | 24.6 | 20.0
  a=Strongly Agree | 31.6 | 25.0
  a=Not Applicable | 3.5 | 1.7
  a=Missing | 5.3 | 11.7
  b=Strongly Disagree | 7.0 | 10.0
  b=Disagree | 14.0 | 8.3
  b=Neutral | 29.8 | 28.3
  b=Agree | 12.3 | 18.3
  b=Strongly Agree | 24.6 | 16.7
  b=Not Applicable | 7.0 | 6.7
  b=Missing | 5.3 | 11.7
  c=Strongly Disagree | 0 | 0
  c=Disagree | 8.8 | 0
  c=Neutral | 29.8 | 53.3
  c=Agree | 26.3 | 18.3
  c=Strongly Agree | 26.3 | 15.0
  c=Not Applicable | 3.5 | 1.7
  c=Missing | 5.3 | 11.7
  d=Strongly Disagree | 12.3 | 20.0
  d=Disagree | 12.3 | 3.3
  d=Neutral | 22.8 | 30.0
  d=Agree | 15.8 | 18.3
  d=Strongly Agree | 28.1 | 15.0
  d=Not Applicable | 3.5 | 1.7
  d=Missing | 5.3 | 11.7
  e=Strongly Disagree | 1.8 | 0
  e=Disagree | 19.3 | 11.7
  e=Neutral | 14.0 | 26.7
  e=Agree | 29.8 | 38.3
  e=Strongly Agree | 26.3 | 10.0
  e=Not Applicable | 3.5 | 1.7
  e=Missing | 5.3 | 11.7
  f=Strongly Disagree | 0 | 1.7
  f=Disagree | 10.5 | 5.0
  f=Neutral | 33.3 | 46.7
  f=Agree | 21.1 | 20.0
  f=Strongly Agree | 26.3 | 8.3
  f=Not Applicable | 3.5 | 6.7
  f=Missing | 5.3 | 11.7
  g=Strongly Disagree | 5.3 | 11.7
  g=Disagree | 5.3 | 1.7
  g=Neutral | 26.3 | 36.7
  g=Agree | 26.3 | 21.7
  g=Strongly Agree | 28.1 | 15.0
  g=Not Applicable | 3.5 | 1.7
  g=Missing | 5.3 | 11.7
  h=Strongly Disagree | 0 | 0
  h=Disagree | 0 | 0
  h=Neutral | 10.5 | 15.0
  h=Agree | 40.4 | 38.3
  h=Strongly Agree | 28.1 | 25.0
  h=Not Applicable | 15.8 | 10.0
  h=Missing | 5.3 | 11.7

6. Secondary Outcome: Percentage of HCPs by Their Response to Perception of Time/Resource Use for Atezolizumab SC and Atezolizumab IV, Assessed Using Questions 3 and 4 of HCPQ - Drug Preparation Area
Description: HCPs who prepared study treatment within the pharmacy/drug preparation area responded at to the following HCPQ-Drug Preparation Area Questions 3 and 4, at Cycle 6 of the Treatment Crossover Period for every participant: "Looking back over the Atezolizumab treatment sessions, please indicate based on your opinion which administration method: Question 3. Was quickest from start to end of preparation to finish of administration (excluding observation period)?; Question 4. Required less resource use for preparation and administration, for example nursing time, facility costs, equipment etc?" The four available response options were: Atezolizumab IV, Atezolizumab SC, No Difference, and Missing. Percentages have been rounded off.
Time Frame: Cycle 6 Day 1 (cycle length= 21 days)
Population: Overall number analyzed included HCPs who completed Questions 3 and 4 of the survey at treatment Cycle 6.
Measure: Number; unit: percentage of HCPs
Arm/Group | Atezolizumab IV/ SC | Atezolizumab SC/ IV
Number analyzed (Participants) | 57 | 60
percentage of HCPs
  Question 3=Atezolizumab SC | 71.9 | 58.3
  Question 3=Atezolizumab IV | 0 | 0
  Question 3=No Difference | 17.5 | 21.7
  Question 3=Missing | 10.5 | 20.0
  Question 4=Atezolizumab SC | 64.9 | 60.0
  Question 4=Atezolizumab IV | 3.5 | 0
  Question 4=No Difference | 21.1 | 20.0
  Question 4=Missing | 10.5 | 20.0

7. Secondary Outcome: Duration of Treatment Administration Activities According to HCPs Response to Perception of Time, Assessed Using Question 1 of HCPQs - Treatment Room
Description: The HCPQ-Treatment Room Question 1 was completed for every participant at each treatment cycle of the Treatment Crossover Period (Cycles 1-6,i.e., 3 cycles of atezolizumab IV followed by 3 cycles of atezolizumab SC/vice versa) by HCPs who administered treatment to the study participants. HCPs responded to following parts of Question 1 that sought to evaluate the amount of time it took to complete activities related to treatment administration: "If new IV access was needed for this cycle of treatment, please indicate what type of IV access was provided (central venous catheter, peripherally inserted central catheter (PICC)/peripheral vein cannulation) & how long (in minutes) this took to set up (only for participants receiving IV treatment)? How long (in minutes) did it take to administer the treatment, i.e. total infusion duration? How long (in minutes) was the participant in the treatment room for in total?" Durations with non-zero HCP responders have been reported here.
Time Frame: Day 1 of Cycles 1 to 6 (cycle length=21 days)
Population: Overall number analyzed included HCPs who completed Question 1 of the survey. For the questions related to IV access, the number analyzed only includes number of HCP responders for participants who required new IV access at a given treatment cycle. The number analyzed included HCPs who completed Question 1 of the survey at the specified treatment cycles. Percentages have been rounded off.
Measure: Median (Full Range); unit: minutes
Arm/Group | Atezolizumab IV/ SC | Atezolizumab SC/ IV
Number analyzed (Participants) | 87 | 86
minutes
  Cycle 1: Duration of Central Venous Catheter set up?: number analyzed (Participants) | 1 | 0
  Cycle 1: Duration of Central Venous Catheter set up? | 5 [5 to 5] |
  Cycle 1: Duration of Peripherally Inserted Central Catheter set up?: number analyzed (Participants) | 3 | 0
  Cycle 1: Duration of Peripherally Inserted Central Catheter set up? | 30.0 [8 to 30] |
  Cycle 1: Duration of Peripheral Vein Cannulation set up?: number analyzed (Participants) | 62 | 0
  Cycle 1: Duration of Peripheral Vein Cannulation set up? | 5.0 [1 to 70] |
  Cycle 1: How Long did it Take to Administer the Treatment?: number analyzed (Participants) | 85 | 86
  Cycle 1: How Long did it Take to Administer the Treatment? | 60.0 [10 to 120] | 8.0 [5 to 75]
  Cycle 1: How Long was the Participant in the Treatment Room in Total?: number analyzed (Participants) | 85 | 86
  Cycle 1: How Long was the Participant in the Treatment Room in Total? | 92.0 [35 to 390] | 55.0 [10 to 260]
  Cycle 2: Duration of Peripherally Inserted Central Catheter set up?: number analyzed (Participants) | 3 | 0
  Cycle 2: Duration of Peripherally Inserted Central Catheter set up? | 30.0 [5 to 35] |
  Cycle 2: Duration of Peripheral Vein Cannulation set up?: number analyzed (Participants) | 52 | 0
  Cycle 2: Duration of Peripheral Vein Cannulation set up? | 5.0 [3.0 to 10.0] |
  Cycle 2: How Long did it Take to Administer the Treatment?: number analyzed (Participants) | 77 | 79
  Cycle 2: How Long did it Take to Administer the Treatment? | 30.0 [13 to 90] | 6.0 [3 to 30]
  Cycle 2: How Long was the Participant in the Treatment Room in Total? | 75.0 [33 to 330] | 41.0 [10 to 238]
  Cycle 3: Duration of Central Venous Catheter set up?: number analyzed (Participants) | 1 | 0
  Cycle 3: Duration of Central Venous Catheter set up? | 61.0 [61 to 61] |
  Cycle 3: Duration of Peripherally Inserted Central Catheter set up?: number analyzed (Participants) | 4 | 0
  Cycle 3: Duration of Peripherally Inserted Central Catheter set up? | 17.5 [5 to 30] |
  Cycle 3: Duration of Peripheral Vein Cannulation set up?: number analyzed (Participants) | 46 | 0
  Cycle 3: Duration of Peripheral Vein Cannulation set up? | 5.0 [1 to 40] |
  Cycle 3: How Long did it Take to Administer the Treatment?: number analyzed (Participants) | 72 | 75
  Cycle 3: How Long did it Take to Administer the Treatment? | 30.0 [20 to 66] | 6.0 [3 to 15]
  Cycle 3: How Long was the Participant in the Treatment Room in Total?: number analyzed (Participants) | 72 | 75
  Cycle 3: How Long was the Participant in the Treatment Room in Total? | 70.0 [35 to 323] | 49.0 [5 to 128]
  Cycle 4: Duration of Central Venous Catheter set up?: number analyzed (Participants) | 0 | 1
  Cycle 4: Duration of Central Venous Catheter set up? |  | 10.0 [10 to 10]
  Cycle 4: Duration of Peripherally Inserted Central Catheter set up?: number analyzed (Participants) | 0 | 5
  Cycle 4: Duration of Peripherally Inserted Central Catheter set up? |  | 30.0 [10.0 to 60.0]
  Cycle 4: Duration of Peripheral Vein Cannulation set up?: number analyzed (Participants) | 0 | 49
  Cycle 4: Duration of Peripheral Vein Cannulation set up? |  | 5.0 [1 to 70]
  Cycle 4: How Long did it Take to Administer the Treatment?: number analyzed (Participants) | 68 | 70
  Cycle 4: How Long did it Take to Administer the Treatment? | 8.0 [5 to 73] | 60.0 [15 to 90]
  Cycle 4: How Long was the Participant in the Treatment Room in Total? | 45.0 [10 to 320] | 97.0 [20 to 360]
  Cycle 5: Duration of Central Venous Catheter set up?: number analyzed (Participants) | 0 | 1
  Cycle 5: Duration of Central Venous Catheter set up? |  | 5.0 [5 to 5]
  Cycle 5: Duration of Peripherally Inserted Central Catheter set up?: number analyzed (Participants) | 0 | 6
  Cycle 5: Duration of Peripherally Inserted Central Catheter set up? |  | 22.5 [7 to 51]
  Cycle 5: Duration of Peripheral Vein Cannulation set up?: number analyzed (Participants) | 0 | 46
  Cycle 5: Duration of Peripheral Vein Cannulation set up? |  | 5.0 [1 to 65]
  Cycle 5: How Long did it Take to Administer the Treatment?: number analyzed (Participants) | 61 | 65
  Cycle 5: How Long did it Take to Administer the Treatment? | 6.0 [1 to 15] | 30.0 [8 to 60]
  Cycle 5: How Long was the Participant in the Treatment Room in Total?: number analyzed (Participants) | 61 | 64
  Cycle 5: How Long was the Participant in the Treatment Room in Total? | 35.0 [8 to 200] | 71.0 [30 to 360]
  Cycle 6: Duration of Peripherally Inserted Central Catheter set up?: number analyzed (Participants) | 0 | 6
  Cycle 6: Duration of Peripherally Inserted Central Catheter set up? |  | 12.5 [5 to 30]
  Cycle 6: Duration of Peripheral Vein Cannulation set up?: number analyzed (Participants) | 0 | 40
  Cycle 6: Duration of Peripheral Vein Cannulation set up? |  | 5.0 [1 to 33]
  Cycle 6: How Long did it Take to Administer the Treatment?: number analyzed (Participants) | 58 | 60
  Cycle 6: How Long did it Take to Administer the Treatment? | 7.0 [1 to 35] | 30.0 [8 to 63]
  Cycle 6: How Long was the Participant in the Treatment Room in Total?: number analyzed (Participants) | 58 | 60
  Cycle 6: How Long was the Participant in the Treatment Room in Total? | 37.5 [9 to 240] | 61.0 [14 to 380]

8. Secondary Outcome: Percentage of HCPs by Their Response to Perception of Impact on Clinical Management and Clinical Efficiency of Atezolizumab SC and IV, Assessed Using Question 2 of HCPQ - Treatment Room
Description: HCPs who administered treatment responded to Question 2: If all IV are switched to SC, please indicate how strongly you agree/disagree with each of following statements: a= Participants will be moved outside of infusion unit to receive SC injections (physician consultation room); b=Atezolizumab SC route will allow more flexible treatment scheduling; c=More participants will be treated in infusion unit; d=Waiting list for any IV treatment at infusion unit will be reduced; e=Staff resources will be re distributed to other departments of the hospital (less staffing required within infusion unit); f=There will still be sufficient interaction time between HCPs & participants (for participant education); g=Staff will spend more time for further professional education/development; h=Staff will dedicate more time to attending to administrative tasks for participants; i=Participants will spend less time in care unit; j=Administration by atezolizumab SC injection is preferred by participants.
Time Frame: Cycle 6 Day 1 (cycle length=21 days)
Population: as for outcome 5
Measure: Number; unit: percentage of HCPs
Arm/Group | Atezolizumab IV/SC | Atezolizumab SC/ IV
Number analyzed (Participants) | 58 | 61
percentage of HCPs
  a=Strongly Disagree | 13.8 | 11.5
  a=Disagree | 15.5 | 23.0
  a=Neutral | 1.7 | 6.6
  a=Agree | 27.6 | 23.0
  a=Strongly Agree | 17.2 | 14.8
  a=Not Applicable | 10.3 | 1.6
  a=Missing | 13.8 | 19.7
  b=Strongly Disagree | 5.3 | 1.6
  b=Disagree | 19.0 | 14.8
  b=Neutral | 10.3 | 21.3
  b=Agree | 22.4 | 21.3
  b=Strongly Agree | 27.6 | 21.3
  b=Not Applicable | 1.7 | 0
  b=Missing | 13.8 | 19.7
  c=Strongly Disagree | 5.2 | 0
  c=Disagree | 15.5 | 16.4
  c=Neutral | 12.1 | 23.0
  c=Agree | 25.9 | 26.2
  c=Strongly Agree | 27.6 | 14.8
  c=Not Applicable | 0 | 0
  c=Missing | 13.8 | 19.7
  d=Strongly Disagree | 6.9 | 1.6
  d=Disagree | 5.2 | 6.6
  d=Neutral | 25.9 | 31.1
  d=Agree | 19.0 | 23.0
  d=Strongly Agree | 27.6 | 18.0
  d=Not Applicable | 1.7 | 0
  d=Missing | 13.8 | 19.7
  e=Strongly Disagree | 13.8 | 11.5
  e=Disagree | 8.6 | 14.8
  e=Neutral | 27.6 | 26.2
  e=Agree | 10.3 | 11.5
  e=Strongly Agree | 19.0 | 13.1
  e=Not Applicable | 6.9 | 3.3
  e=Missing | 13.8 | 19.7
  f=Strongly Disagree | 0 | 0
  f=Disagree | 17.2 | 11.5
  f=Neutral | 17.2 | 32.8
  f=Agree | 22.4 | 16.4
  f=Strongly Agree | 29.3 | 19.7
  f=Not Applicable | 0 | 0
  f=Missing | 13.8 | 19.7
  g=Strongly Disagree | 6.9 | 1.6
  g=Disagree | 12.1 | 11.5
  g=Neutral | 27.6 | 27.9
  g=Agree | 13.8 | 24.6
  g=Strongly Agree | 25.9 | 14.8
  g=Not Applicable | 0 | 0
  g=Missing | 13.8 | 19.7
  h=Strongly Disagree | 6.9 | 0
  h=Disagree | 17.2 | 24.6
  h=Neutral | 15.5 | 13.1
  h=Agree | 24.1 | 29.5
  h=Strongly Agree | 20.7 | 13.1
  h=Not Applicable | 1.7 | 0
  h=Missing | 13.8 | 19.7
  i=Strongly Disagree | 1.7 | 1.6
  i=Disagree | 5.2 | 4.9
  i=Neutral | 8.6 | 14.8
  i=Agree | 37.9 | 27.9
  i=Strongly Agree | 32.8 | 31.1
  i=Not Applicable | 0 | 0
  i=Missing | 13.8 | 19.7
  j=Strongly Disagree | 1.7 | 1.6
  j=Disagree | 0 | 3.3
  j=Neutral | 20.7 | 21.3
  j=Agree | 31.0 | 27.9
  j=Strongly Agree | 31.0 | 26.2
  j=Not Applicable | 1.7 | 0
  j=Missing | 13.8 | 19.7

9. Secondary Outcome: Percentage of HCPs by Their Response to Perception of Time/Resource Use and Convenience for Atezolizumab SC and Atezolizumab IV, Assessed Using Questions 3 to 7 of HCPQ - Treatment Room
Description: HCPs who administered study treatment responded at Cycle 6 of the Treatment Crossover Period to the following HCPQ-treatment room Questions 3 to 7: "Looking back over the atezolizumab treatment sessions, please indicate based on your opinion which administration method: Question 3. Which method was most convenient for the participant? Question 4. Which method was best for optimizing participant care in your center? Question 5. Which method took the least time from start to finish of administration? Question 6. Which method required the least resource use for administration? Question 7. Which method was preferred by participants?" The five available response options were: Atezolizumab SC, Atezolizumab IV, No Difference, Unsure and Missing. Percentages have been rounded off.
Time Frame: Cycle 6 Day 1 (cycle length=21 days)
Population: Overall number analyzed included HCPs who completed Questions 3 to 7 of the survey at treatment Cycle 6.
Measure: Number; unit: percentage of HCPs
Arm/Group | Atezolizumab IV/ SC | Atezolizumab SC/ IV
Number analyzed (Participants) | 58 | 61
percentage of HCPs
  Q3=Atezolizumab SC | 72.4 | 63.9
  Q3=Atezolizumab IV | 5.2 | 10.1
  Q3=No Difference | 6.9 | 8.4
  Q3=Unsure | 1.7 | 3.3
  Q3= Missing | 13.8 | 14.4
  Q4=Atezolizumab SC | 55.2 | 39.3
  Q4=Atezolizumab IV | 6.9 | 1.5
  Q4=No Difference | 20.7 | 31.1
  Q4=Unsure | 3.4 | 1.6
  Q4=Missing | 13.8 | 16.4
  Q5=Atezolizumab SC | 67.2 | 52.5
  Q5=Atezolizumab IV | 0 | 3.3
  Q5=No Difference | 17.2 | 27.9
  Q5=Unsure | 0 | 0
  Q5=Missing | 15.5 | 16.4
  Q6=Atezolizumab SC | 63.8 | 50.8
  Q6=Atezolizumab IV | 3.4 | 1.6
  Q6=No Difference | 19.0 | 31.1
  Q6=Unsure | 0 | 0
  Q6=Missing | 13.8 | 16.4
  Q7=Atezolizumab SC | 63.8 | 52.5
  Q7=Atezolizumab IV | 10.3 | 14.8
  Q7=No Difference | 3.4 | 1.6
  Q7=Unsure | 8.6 | 14.8
  Q7=Missing | 13.8 | 16.4

10. Secondary Outcome: Percentage of HCPs by Their Response to Perception of Time/Resource Use and Convenience for Atezolizumab SC and Atezolizumab IV, Assessed Using Questions 8 of HCPQ - Treatment Room
Description: HCPs who administered study treatment responded at Cycle 6 of the treatment Cross-over Period to the following HCPQ-treatment room Question 8: How frequently would you offer or recommend atezolizumab SC administration to your participants in the future? The four available response options were Always, Sometimes, Never and Missing. Percentages have been rounded off.
Time Frame: Cycle 6 Day 1 (cycle length= 21 days)
Population: Overall number analyzed included HCPs who completed Question 8 of the survey at treatment Cycle 6.
Measure: Number; unit: percentage of HCPs
Arm/Group | Atezolizumab IV/ SC | Atezolizumab SC/ IV
Number analyzed (Participants) | 58 | 61
percentage of HCPs
  Question 8=Always | 41.4 | 31.1
  Question 8=Sometimes | 34.5 | 37.7
  Question 8=Never | 10.3 | 14.8
  Question 8=Missing | 13.8 | 16.4

11. Secondary Outcome: Change From Baseline Over Time in Physical Functioning Scale Score as Assessed by European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC-QLQ-C30)
Description: EORTC QLQ-C30 consists of 30 questions that assess five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), global health status (GHS) and quality of life (QoL), and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) with a recall period of the previous week. Scale scores can be obtained for the multi-item scales. The functioning items are scored on a 4-point scale (1=Not at All to 4=Very Much). Scores are linearly transformed on a scale of 0 to 100, with a high score indicating better functioning. EORTC QLQ-C30 data was scored according to the EORTC scoring manual v3.0. In the event of incomplete data, if more than 50% of the constituent items were completed, a pro-rated score was computed. For subscales with less than 50% of the items completed, the subscale was considered as missing.
Time Frame: Baseline, Day 1 of Cycles 3, 6, 7, 10, 13, 16 and End of Treatment (up to approximately 2.2 years)
Population: FAS included all randomized participants. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Continuation Atezolizumab IV: After 6 cycles of Crossover Period, participants were given an option to choose between IV or SC administration of atezolizumab for the Treatment Continuation Period. Participants in this arm chose to continue treatment with atezolizumab IV, 1200 mg Q3W up to Cycle 16 for participants with early-stage NSCLC or until loss of clinical benefit for participants with advanced NSCLC.
- Continuation Atezolizumab SC: After 6 cycles of Crossover Period, participants were given an option to choose between IV or SC administration of atezolizumab for the Treatment Continuation Period. Participants in this arm chose to continue treatment with atezolizumab SC, 1875 mg Q3W up to Cycle 16 for participants with early-stage NSCLC or until loss of clinical benefit for participants with advanced NSCLC.
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Number analyzed (Participants) | 88 | 85 | 24 | 82
score on a scale
  Baseline: number analyzed (Participants) | 88 | 85 | 0 | 0
  Baseline | 75.00 (19.79) | 72.09 (20.10) |  |
  Change at Cycle 3 Day 1: number analyzed (Participants) | 72 | 75 | 0 | 0
  Change at Cycle 3 Day 1 | -0.46 (19.62) | -2.01 (16.00) |  |
  Change at Cycle 6 Day 1: number analyzed (Participants) | 58 | 61 | 0 | 0
  Change at Cycle 6 Day 1 | 0.00 (16.19) | -1.60 (16.74) |  |
  Change at Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 24 | 76
  Change at Cycle 7 Day 1 |  |  | -2.22 (13.85) | 0.03 (15.39)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 22 | 82
  Change at Cycle 10 Day 1 |  |  | 0.91 (19.55) | 2.06 (16.64)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 17 | 73
  Change at Cycle 13 Day 1 |  |  | -5.10 (19.93) | -0.43 (17.98)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 14 | 67
  Change at Cycle 16 Day 1 |  |  | 0.48 (16.22) | 1.03 (15.77)
  Change at End of Treatment: number analyzed (Participants) | 12 | 10 | 24 | 76
  Change at End of Treatment | -13.75 (28.39) | -14.67 (25.49) | -8.06 (21.26) | -3.92 (21.67)

12. Secondary Outcome: Change From Baseline Over Time in Role Functioning Scale Score as Assessed by EORTC-QLQ-C30
Description: EORTC QLQ-C30 consists of 30 questions that assess five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), GHS and QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) with a recall period of the previous week. Scale scores can be obtained for the multi-item scales. The functioning items are scored on a 4-point scale (1=Not at All to 4=Very Much). Scores are linearly transformed on a scale of 0 to 100, with a high score indicating better functioning. EORTC QLQ-C30 data was scored according to the EORTC scoring manual v3.0. In the event of incomplete data, if more than 50% of the constituent items were completed, a pro-rated score was computed. For subscales with less than 50% of the items completed, the subscale was considered as missing.
Time Frame: Baseline, Day 1 of Cycles 3, 6, 7, 10, 13, 16 and End of Treatment (up to approximately 2.2 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Number analyzed (Participants) | 88 | 85 | 24 | 82
score on a scale
  Baseline: number analyzed (Participants) | 88 | 85 | 0 | 0
  Baseline | 77.46 (25.15) | 73.73 (27.86) |  |
  Change at Cycle 3 Day 1: number analyzed (Participants) | 72 | 75 | 0 | 0
  Change at Cycle 3 Day 1 | 1.16 (29.25) | -1.33 (21.88) |  |
  Change at Cycle 6 Day 1: number analyzed (Participants) | 58 | 61 | 0 | 0
  Change at Cycle 6 Day 1 | -2.01 (26.13) | -1.64 (24.10) |  |
  Change at Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 24 | 77
  Change at Cycle 7 Day 1 |  |  | -8.33 (18.39) | -5.41 (26.00)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 22 | 82
  Change at Cycle 10 Day 1 |  |  | -6.82 (23.94) | -2.03 (24.20)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 17 | 73
  Change at Cycle 13 Day 1 |  |  | -6.86 (21.29) | -1.60 (26.52)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 14 | 67
  Change at Cycle 16 Day 1 |  |  | -2.38 (14.41) | -2.74 (26.84)
  Change at End of Treatment: number analyzed (Participants) | 12 | 10 | 24 | 77
  Change at End of Treatment | -16.67 (43.81) | -15.00 (24.15) | -9.72 (24.04) | -8.01 (25.88)

13. Secondary Outcome: Change From Baseline Over Time in Emotional Functioning Scale Score as Assessed by EORTC-QLQ-C30
Description: as for outcome 12
Time Frame: Baseline, Day 1 of Cycles 3, 6, 7, 10, 13, 16 and End of Treatment (up to approximately 2.2 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Number analyzed (Participants) | 88 | 85 | 24 | 82
score on a scale
  Baseline: number analyzed (Participants) | 88 | 85 | 0 | 0
  Baseline | 79.48 (22.43) | 75.98 (23.44) |  |
  Change at Cycle 3 Day 1: number analyzed (Participants) | 72 | 75 | 0 | 0
  Change at Cycle 3 Day 1 | 2.62 (20.52) | 0.89 (16.47) |  |
  Change at Cycle 6 Day 1: number analyzed (Participants) | 58 | 61 | 0 | 0
  Change at Cycle 6 Day 1 | 0.77 (17.68) | 4.10 (23.30) |  |
  Change at Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 24 | 77
  Change at Cycle 7 Day 1 |  |  | -3.47 (22.64) | 2.56 (15.84)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 22 | 82
  Change at Cycle 10 Day 1 |  |  | -3.03 (26.92) | 4.37 (16.91)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 17 | 73
  Change at Cycle 13 Day 1 |  |  | 0.98 (22.61) | 3.46 (19.00)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 14 | 67
  Change at Cycle 16 Day 1 |  |  | -2.98 (23.02) | 0.37 (17.49)
  Change at End of Treatment: number analyzed (Participants) | 12 | 10 | 24 | 77
  Change at End of Treatment | -6.71 (16.98) | -6.67 (21.08) | -8.33 (28.45) | -5.05 (18.16)

14. Secondary Outcome: Change From Baseline Over Time in Cognitive Functioning Scale Score as Assessed by EORTC-QLQ-C30
Description: as for outcome 12
Time Frame: Baseline, Day 1 of Cycles 3, 6, 7, 10, 13, 16 and End of Treatment (up to approximately 2.2 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Number analyzed (Participants) | 88 | 85 | 24 | 82
score on a scale
  Baseline: number analyzed (Participants) | 88 | 85 | 0 | 0
  Baseline | 87.31 (21.74) | 85.69 (19.78) |  |
  Change at Cycle 3 Day 1: number analyzed (Participants) | 72 | 75 | 0 | 0
  Change at Cycle 3 Day 1 | 2.31 (17.31) | -5.56 (19.05) |  |
  Change at Cycle 6 Day 1: number analyzed (Participants) | 58 | 61 | 0 | 0
  Change at Cycle 6 Day 1 | -5.75 (18.87) | -1.09 (20.15) |  |
  Change at Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 24 | 77
  Change at Cycle 7 Day 1 |  |  | -4.17 (13.23) | -2.16 (19.37)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 22 | 82
  Change at Cycle 10 Day 1 |  |  | -5.30 (11.94) | -0.41 (17.76)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 17 | 73
  Change at Cycle 13 Day 1 |  |  | -11.76 (21.86) | -1.14 (21.21)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 14 | 67
  Change at Cycle 16 Day 1 |  |  | -7.14 (12.60) | -2.99 (21.11)
  Change at End of Treatment: number analyzed (Participants) | 12 | 10 | 24 | 77
  Change at End of Treatment | -6.94 (25.08) | 3.33 (17.21) | -5.56 (23.40) | -7.36 (22.70)

15. Secondary Outcome: Change From Baseline Over Time in Social Functioning Scale Score as Assessed by EORTC-QLQ-C30
Description: as for outcome 12
Time Frame: Baseline, Day 1 of Cycles 3, 6, 7, 10, 13, 16 and End of Treatment (up to approximately 2.2 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Number analyzed (Participants) | 88 | 85 | 24 | 82
score on a scale
  Baseline: number analyzed (Participants) | 88 | 85 | 0 | 0
  Baseline | 82.95 (23.02) | 82.35 (22.76) |  |
  Change at Cycle 3 Day 1: number analyzed (Participants) | 72 | 75 | 0 | 0
  Change at Cycle 3 Day 1 | 3.70 (23.61) | -3.56 (21.10) |  |
  Change at Cycle 6 Day 1: number analyzed (Participants) | 58 | 61 | 0 | 0
  Change at Cycle 6 Day 1 | -2.87 (24.81) | -1.91 (22.38) |  |
  Change at Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 24 | 77
  Change at Cycle 7 Day 1 |  |  | -6.25 (27.72) | 0.22 (21.71)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 22 | 82
  Change at Cycle 10 Day 1 |  |  | -3.79 (27.18) | -0.20 (25.32)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 17 | 73
  Change at Cycle 13 Day 1 |  |  | -3.92 (17.21) | -0.46 (23.57)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 14 | 67
  Change at Cycle 16 Day 1 |  |  | -5.95 (24.11) | 0.50 (19.67)
  Change at End of Treatment: number analyzed (Participants) | 12 | 10 | 24 | 77
  Change at End of Treatment | -12.50 (46.13) | -15.00 (29.87) | -15.28 (24.53) | -4.98 (27.84)

16. Secondary Outcome: Change From Baseline Over Time in Fatigue Scale Score as Assessed by EORTC-QLQ-C30
Description: EORTC QLQ-C30 consists of 30 questions that assess five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), GHS and QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) with a recall period of the previous week. Scale scores can be obtained for the multi-item scales. The symptom items are scored on a 4-point scale (1=Not at All to 4=Very Much). Scores are linearly transformed on a scale of 0 to 100, with a high score indicating worst symptoms. EORTC QLQ-C30 data was scored according to the EORTC scoring manual v3.0. In the event of incomplete data, if more than 50% of the constituent items were completed, a pro-rated score was computed. For subscales with less than 50% of the items completed, the subscale was considered as missing.
Time Frame: Baseline, Day 1 of Cycles 3, 6, 7, 10, 13, 16 and End of Treatment (up to approximately 2.2 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Number analyzed (Participants) | 88 | 85 | 24 | 82
score on a scale
  Baseline: number analyzed (Participants) | 88 | 85 | 0 | 0
  Baseline | 30.81 (25.81) | 36.08 (26.33) |  |
  Change at Cycle 3 Day 1: number analyzed (Participants) | 72 | 75 | 0 | 0
  Change at Cycle 3 Day 1 | 0.15 (26.67) | -1.63 (20.32) |  |
  Change at Cycle 6 Day 1: number analyzed (Participants) | 58 | 61 | 0 | 0
  Change at Cycle 6 Day 1 | 4.41 (25.06) | 1.46 (21.13) |  |
  Change at Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 24 | 77
  Change at Cycle 7 Day 1 |  |  | 2.78 (18.02) | 1.59 (23.27)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 22 | 82
  Change at Cycle 10 Day 1 |  |  | 3.03 (21.74) | -0.14 (21.63)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 17 | 73
  Change at Cycle 13 Day 1 |  |  | 4.58 (15.24) | 3.96 (26.02)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 14 | 67
  Change at Cycle 16 Day 1 |  |  | 5.56 (20.32) | 1.00 (26.64)
  Change at End of Treatment: number analyzed (Participants) | 12 | 10 | 24 | 77
  Change at End of Treatment | 6.48 (24.37) | 4.44 (24.68) | 1.39 (27.86) | 7.65 (24.13)

17. Secondary Outcome: Change From Baseline Over Time in Nausea and Vomiting Scale Score as Assessed by EORTC-QLQ-C30
Description: as for outcome 16
Time Frame: Baseline, Day 1 of Cycles 3, 6, 7, 10, 13, 16 and End of Treatment (up to approximately 2.2 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Number analyzed (Participants) | 88 | 85 | 24 | 82
score on a scale
  Baseline: number analyzed (Participants) | 88 | 85 | 0 | 0
  Baseline | 5.30 (13.50) | 5.88 (14.48) |  |
  Change at Cycle 3 Day 1: number analyzed (Participants) | 72 | 75 | 0 | 0
  Change at Cycle 3 Day 1 | 2.31 (15.65) | 1.56 (18.21) |  |
  Change at Cycle 6 Day 1: number analyzed (Participants) | 58 | 61 | 0 | 0
  Change at Cycle 6 Day 1 | 2.01 (12.90) | 3.01 (14.11) |  |
  Change at Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 24 | 77
  Change at Cycle 7 Day 1 |  |  | 4.86 (9.17) | -0.65 (9.15)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 22 | 82
  Change at Cycle 10 Day 1 |  |  | 3.79 (10.20) | 1.02 (9.57)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 17 | 73
  Change at Cycle 13 Day 1 |  |  | 0.98 (4.04) | 0.46 (14.16)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 14 | 67
  Change at Cycle 16 Day 1 |  |  | 1.19 (4.45) | 0.75 (13.11)
  Change at End of Treatment: number analyzed (Participants) | 11 | 10 | 24 | 77
  Change at End of Treatment | -3.03 (16.36) | 6.67 (23.83) | 6.94 (18.33) | 1.73 (12.56)

18. Secondary Outcome: Change From Baseline Over Time in Pain Scale Score as Assessed by EORTC-QLQ-C30
Description: as for outcome 16
Time Frame: Baseline, Day 1 of Cycles 3, 6, 7, 10, 13, 16 and End of Treatment (up to approximately 2.2 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Number analyzed (Participants) | 88 | 85 | 24 | 82
score on a scale
  Baseline: number analyzed (Participants) | 88 | 85 | 0 | 0
  Baseline | 22.16 (25.23) | 29.22 (30.74) |  |
  Change at Cycle 3 Day 1: number analyzed (Participants) | 72 | 75 | 0 | 0
  Change at Cycle 3 Day 1 | 0.93 (22.88) | -3.56 (26.47) |  |
  Change at Cycle 6 Day 1: number analyzed (Participants) | 58 | 61 | 0 | 0
  Change at Cycle 6 Day 1 | 4.02 (23.22) | -1.09 (25.43) |  |
  Change at Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 24 | 77
  Change at Cycle 7 Day 1 |  |  | 4.17 (28.34) | 1.52 (28.89)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 22 | 82
  Change at Cycle 10 Day 1 |  |  | 3.79 (32.50) | -1.22 (26.42)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 17 | 73
  Change at Cycle 13 Day 1 |  |  | 7.84 (35.90) | 1.14 (25.81)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 14 | 67
  Change at Cycle 16 Day 1 |  |  | 4.76 (32.31) | 1.24 (28.32)
  Change at End of Treatment: number analyzed (Participants) | 12 | 10 | 24 | 77
  Change at End of Treatment | 12.50 (43.30) | -10.00 (28.54) | 18.06 (33.66) | 6.28 (30.35)

19. Secondary Outcome: Change From Baseline Over Time in Dyspnoea Scale Score as Assessed by EORTC-QLQ-C30
Description: EORTC QLQ-C30 consists of 30 questions that assess five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), GHS and QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) with a recall period of the previous week. Scale scores can be obtained for the multi-item scales. The dyspnoea scale items are scored on a 4-point scale (1=Not at All to 4=Very Much). Scores are linearly transformed on a scale of 0 to 100, with a high score the scale indicating worst symptoms. EORTC QLQ-C30 data was scored according to the EORTC scoring manual v3.0. In the event of incomplete data, if more than 50% of the constituent items were completed, a pro-rated score was computed. For subscales with less than 50% of the items completed, the subscale was considered as missing.
Time Frame: Baseline, Day 1 of Cycles 3, 6, 7, 10, 13, 16 and End of Treatment (up to approximately 2.2 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Number analyzed (Participants) | 88 | 85 | 24 | 82
score on a scale
  Baseline: number analyzed (Participants) | 88 | 85 | 0 | 0
  Baseline | 25.38 (26.26) | 30.59 (30.52) |  |
  Change at Cycle 3 Day 1: number analyzed (Participants) | 72 | 75 | 0 | 0
  Change at Cycle 3 Day 1 | 5.09 (26.63) | 0.89 (26.83) |  |
  Change at Cycle 6 Day 1: number analyzed (Participants) | 58 | 61 | 0 | 0
  Change at Cycle 6 Day 1 | -0.57 (22.07) | -2.73 (31.80) |  |
  Change at Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 24 | 77
  Change at Cycle 7 Day 1 |  |  | 4.17 (31.57) | -3.03 (27.14)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 22 | 82
  Change at Cycle 10 Day 1 |  |  | 3.03 (25.01) | -5.28 (25.37)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 17 | 73
  Change at Cycle 13 Day 1 |  |  | 0.00 (28.87) | 0.00 (24.22)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 14 | 67
  Change at Cycle 16 Day 1 |  |  | 0.00 (29.24) | -4.48 (26.52)
  Change at End of Treatment: number analyzed (Participants) | 12 | 10 | 24 | 77
  Change at End of Treatment | 8.33 (15.08) | 16.67 (28.33) | 4.17 (31.57) | 2.60 (26.36)

20. Secondary Outcome: Change From Baseline Over Time in Insomnia Scale Score as Assessed by EORTC-QLQ-C30
Description: EORTC QLQ-C30 consists of 30 questions that assess five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), GHS and QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) with a recall period of the previous week. Scale scores can be obtained for the multi-item scales. The insomnia scale items are scored on a 4-point scale (1=Not at All to 4=Very Much). Scores are linearly transformed on a scale of 0 to 100, with a high score on the scale indicating worst symptoms. EORTC QLQ-C30 data was scored according to the EORTC scoring manual v3.0. In the event of incomplete data, if more than 50% of the constituent items were completed, a pro-rated score was computed. For subscales with less than 50% of the items completed, the subscale was considered as missing.
Time Frame: Baseline, Day 1 of Cycles 3, 6, 7, 10, 13, 16 and End of Treatment (up to approximately 2.2 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Number analyzed (Participants) | 88 | 85 | 24 | 82
score on a scale
  Baseline: number analyzed (Participants) | 88 | 85 | 0 | 0
  Baseline | 23.11 (27.85) | 28.63 (31.77) |  |
  Change at Cycle 3 Day 1: number analyzed (Participants) | 72 | 75 | 0 | 0
  Change at Cycle 3 Day 1 | 0.46 (26.53) | -0.44 (20.13) |  |
  Change at Cycle 6 Day 1: number analyzed (Participants) | 58 | 61 | 0 | 0
  Change at Cycle 6 Day 1 | 0.57 (23.77) | 2.19 (27.13) |  |
  Change at Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 24 | 77
  Change at Cycle 7 Day 1 |  |  | 15.28 (32.57) | 2.16 (23.78)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 22 | 82
  Change at Cycle 10 Day 1 |  |  | 6.06 (24.42) | 2.44 (25.00)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 17 | 73
  Change at Cycle 13 Day 1 |  |  | 15.69 (20.81) | 1.37 (25.72)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 14 | 67
  Change at Cycle 16 Day 1 |  |  | 0.00 (13.07) | 3.98 (22.11)
  Change at End of Treatment: number analyzed (Participants) | 12 | 10 | 24 | 77
  Change at End of Treatment | -2.78 (17.16) | -13.33 (35.83) | 4.17 (38.46) | 3.90 (25.35)

21. Secondary Outcome: Change From Baseline Over Time in Appetite Loss Scale Score as Assessed by EORTC-QLQ-C30
Description: EORTC QLQ-C30 consists of 30 questions that assess five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), GHS and QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) with a recall period of the previous week. Scale scores can be obtained for the multi-item scales. The appetite loss scale items are scored on a 4-point scale (1=Not at All to 4=Very Much). Scores are linearly transformed on a scale of 0 to 100, with a high score on the scale indicating worst symptoms. EORTC QLQ-C30 data was scored according to the EORTC scoring manual v3.0. In the event of incomplete data, if more than 50% of the constituent items were completed, a pro-rated score was computed. For subscales with less than 50% of the items completed, the subscale was considered as missing.
Time Frame: Baseline, Day 1 of Cycles 3, 6, 7, 10, 13, 16 and End of Treatment (up to approximately 2.2 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Number analyzed (Participants) | 88 | 85 | 24 | 82
score on a scale
  Baseline: number analyzed (Participants) | 88 | 85 | 0 | 0
  Baseline | 16.67 (28.14) | 21.96 (28.43) |  |
  Change at Cycle 3 Day 1: number analyzed (Participants) | 72 | 75 | 0 | 0
  Change at Cycle 3 Day 1 | 2.31 (32.30) | 2.22 (23.46) |  |
  Change at Cycle 6 Day 1: number analyzed (Participants) | 58 | 61 | 0 | 0
  Change at Cycle 6 Day 1 | 2.87 (30.13) | -2.19 (26.44) |  |
  Change at Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 24 | 77
  Change at Cycle 7 Day 1 |  |  | 4.17 (30.00) | -3.03 (27.14)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 22 | 82
  Change at Cycle 10 Day 1 |  |  | 6.06 (35.09) | -2.03 (25.31)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 17 | 73
  Change at Cycle 13 Day 1 |  |  | -1.96 (18.52) | -0.46 (26.35)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 14 | 67
  Change at Cycle 16 Day 1 |  |  | 0.00 (13.07) | 0.00 (25.29)
  Change at End of Treatment: number analyzed (Participants) | 11 | 10 | 24 | 76
  Change at End of Treatment | -6.06 (25.03) | 3.33 (36.68) | 0.00 (31.08) | 2.63 (25.97)

22. Secondary Outcome: Change From Baseline Over Time in Constipation Scale Score as Assessed by EORTC-QLQ-C30
Description: EORTC QLQ-C30 consists of 30 questions that assess five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), GHS and QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) with a recall period of the previous week. Scale scores can be obtained for the multi-item scales. The constipation scale items are scored on a 4-point scale (1=Not at All to 4=Very Much). Scores are linearly transformed on a scale of 0 to 100, with a high score on the scale indicating worst symptoms. EORTC QLQ-C30 data was scored according to the EORTC scoring manual v3.0. In the event of incomplete data, if more than 50% of the constituent items were completed, a pro-rated score was computed. For subscales with less than 50% of the items completed, the subscale was considered as missing.
Time Frame: Baseline, Day 1 of Cycles 3, 6, 7, 10, 13, 16 and End of Treatment (up to approximately 2.2 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Number analyzed (Participants) | 88 | 85 | 24 | 82
score on a scale
  Baseline: number analyzed (Participants) | 88 | 85 | 0 | 0
  Baseline | 19.32 (30.63) | 21.96 (33.55) |  |
  Change at Cycle 3 Day 1: number analyzed (Participants) | 72 | 75 | 0 | 0
  Change at Cycle 3 Day 1 | 0.00 (29.07) | -2.67 (32.77) |  |
  Change at Cycle 6 Day 1: number analyzed (Participants) | 58 | 61 | 0 | 0
  Change at Cycle 6 Day 1 | -4.60 (28.92) | -3.28 (30.25) |  |
  Change at Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 24 | 77
  Change at Cycle 7 Day 1 |  |  | -4.17 (20.41) | -9.52 (34.98)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 22 | 82
  Change at Cycle 10 Day 1 |  |  | -3.03 (25.01) | -6.10 (30.60)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 17 | 73
  Change at Cycle 13 Day 1 |  |  | -1.96 (21.96) | -4.11 (29.37)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 14 | 67
  Change at Cycle 16 Day 1 |  |  | -4.76 (17.82) | -1.00 (32.29)
  Change at End of Treatment: number analyzed (Participants) | 11 | 10 | 24 | 77
  Change at End of Treatment | -12.12 (45.39) | 16.67 (39.28) | 1.39 (23.01) | -3.46 (35.29)

23. Secondary Outcome: Change From Baseline Over Time in Diarrhoea Scale Score as Assessed by EORTC-QLQ-C30
Description: EORTC QLQ-C30 consists of 30 questions that assess five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), GHS and QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) with a recall period of the previous week. Scale scores can be obtained for the multi-item scales. The diarrhoea scale items are scored on a 4-point scale (1=Not at All to 4=Very Much). Scores are linearly transformed on a scale of 0 to 100, with a high score on the scale indicating worst symptoms. EORTC QLQ-C30 data was scored according to the EORTC scoring manual v3.0. In the event of incomplete data, if more than 50% of the constituent items were completed, a pro-rated score was computed. For subscales with less than 50% of the items completed, the subscale was considered as missing.
Time Frame: Baseline, Day 1 of Cycles 3, 6, 7, 10, 13, 16 and End of Treatment (up to approximately 2.2 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Number analyzed (Participants) | 88 | 85 | 24 | 82
score on a scale
  Baseline: number analyzed (Participants) | 88 | 85 | 0 | 0
  Baseline | 5.68 (15.35) | 7.06 (15.51) |  |
  Change at Cycle 3 Day 1: number analyzed (Participants) | 72 | 75 | 0 | 0
  Change at Cycle 3 Day 1 | 0.93 (18.53) | 2.22 (18.45) |  |
  Change at Cycle 6 Day 1: number analyzed (Participants) | 58 | 61 | 0 | 0
  Change at Cycle 6 Day 1 | -2.30 (17.51) | 3.28 (21.69) |  |
  Change at Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 24 | 77
  Change at Cycle 7 Day 1 |  |  | 2.78 (16.79) | -1.30 (19.82)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 22 | 82
  Change at Cycle 10 Day 1 |  |  | 4.55 (18.67) | 2.03 (19.14)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 17 | 73
  Change at Cycle 13 Day 1 |  |  | 9.80 (34.89) | -1.83 (16.56)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 14 | 67
  Change at Cycle 16 Day 1 |  |  | 9.52 (30.46) | 0.50 (22.09)
  Change at End of Treatment: number analyzed (Participants) | 12 | 10 | 24 | 77
  Change at End of Treatment | -5.56 (19.25) | -13.33 (23.31) | 5.56 (27.22) | -0.43 (20.59)

24. Secondary Outcome: Change From Baseline Over Time in Financial Difficulties Scale Score as Assessed by EORTC-QLQ-C30
Description: EORTC QLQ-C30 consists of 30 questions that assess five aspects of participant functioning (physical, emotional, role, cognitive, and social), three symptom scales (fatigue, nausea and vomiting, and pain), GHS and QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties) with a recall period of the previous week. Scale scores can be obtained for the multi-item scales. The financial difficulties scale items are scored on a 4-point scale (1=Not at All to 4=Very Much). Scores are linearly transformed on a scale of 0 to 100, with a high score on the scale indicating worst functioning. EORTC QLQ-C30 data was scored according to the EORTC scoring manual v3.0. In the event of incomplete data, if more than 50% of the constituent items were completed, a pro-rated score was computed. For subscales with less than 50% of the items completed, the subscale was considered as missing.
Time Frame: Baseline, Day 1 of Cycles 3, 6, 7, 10, 13, 16 and End of Treatment (up to approximately 2.2 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Number analyzed (Participants) | 87 | 85 | 24 | 81
score on a scale
  Baseline: number analyzed (Participants) | 87 | 85 | 0 | 0
  Baseline | 13.79 (25.19) | 20.39 (31.33) |  |
  Change at Cycle 3 Day 1: number analyzed (Participants) | 71 | 75 | 0 | 0
  Change at Cycle 3 Day 1 | 7.98 (27.87) | -1.33 (23.53) |  |
  Change at Cycle 6 Day 1: number analyzed (Participants) | 57 | 61 | 0 | 0
  Change at Cycle 6 Day 1 | 11.11 (32.33) | 0.00 (25.09) |  |
  Change at Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 24 | 76
  Change at Cycle 7 Day 1 |  |  | 0.00 (17.03) | -0.44 (28.54)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 22 | 81
  Change at Cycle 10 Day 1 |  |  | 0.00 (14.55) | 1.65 (27.34)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 17 | 71
  Change at Cycle 13 Day 1 |  |  | -1.96 (14.29) | 2.35 (28.35)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 14 | 67
  Change at Cycle 16 Day 1 |  |  | -2.38 (8.91) | 5.47 (26.33)
  Change at End of Treatment: number analyzed (Participants) | 11 | 10 | 24 | 76
  Change at End of Treatment | 24.24 (44.95) | 0.00 (35.14) | -1.39 (20.80) | 5.70 (29.51)

25. Secondary Outcome: Change From Baseline Over Time in Health-related Quality of Life (HRQoL) Score as Assessed by GHS/QoL Scale of the EORTC-QLQ-C30
Description: EORTC QLQ-C30 consists of 30 questions that assess participant functioning (physical, emotional, role, cognitive, and social), symptom scales (fatigue, nausea and vomiting, pain), global health/ QoL, and six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Change in HRQoL was assessed using participant responses to questions regarding Global Health Status (Q29: GHS; "How would you rate your overall health during the past week?") and QoL (Q30: QoL; "How would you rate your overall quality of life during the past week?") and were scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized. Scores range from 0-100. A higher score indicates a better outcome.
Time Frame: Baseline, Day 1 of Cycles 3, 6, 7, 10, 13, 16 and End of Treatment (up to approximately 2.2 years)
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Crossover Atezolizumab IV/SC | Crossover Atezolizumab SC/IV | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Number analyzed (Participants) | 87 | 85 | 24 | 82
score on a scale
  Baseline: number analyzed (Participants) | 87 | 85 | 0 | 0
  Baseline | 67.05 (19.97) | 64.80 (21.45) |  |
  Change at Cycle 3 Day 1: number analyzed (Participants) | 71 | 75 | 0 | 0
  Change at Cycle 3 Day 1 | 0.12 (22.95) | -0.22 (18.43) |  |
  Change at Cycle 6 Day 1: number analyzed (Participants) | 57 | 61 | 0 | 0
  Change at Cycle 6 Day 1 | -2.49 (18.83) | -0.27 (22.26) |  |
  Change at Cycle 7 Day 1: number analyzed (Participants) | 0 | 0 | 24 | 77
  Change at Cycle 7 Day 1 |  |  | -2.08 (19.85) | 1.84 (19.94)
  Change at Cycle 10 Day 1: number analyzed (Participants) | 0 | 0 | 22 | 82
  Change at Cycle 10 Day 1 |  |  | -3.79 (16.21) | 1.73 (17.65)
  Change at Cycle 13 Day 1: number analyzed (Participants) | 0 | 0 | 17 | 73
  Change at Cycle 13 Day 1 |  |  | -5.39 (15.29) | 0.23 (19.24)
  Change at Cycle 16 Day 1: number analyzed (Participants) | 0 | 0 | 14 | 67
  Change at Cycle 16 Day 1 |  |  | -7.74 (18.33) | 3.23 (21.07)
  Change at End of Treatment: number analyzed (Participants) | 11 | 10 | 24 | 77
  Change at End of Treatment | -28.79 (26.71) | -11.67 (19.72) | -13.54 (25.40) | -4.76 (22.56)

26. Secondary Outcome: Percentage of Participants With Ongoing Clinical Benefit
Description: Participants were assessed for clinical benefit at every tumour assessment visit, which was conducted as per the local standard of care. Percentages have been rounded off.
Time Frame: Up to Cycle 16 (cycle length= 21 days)
Population: FAS included all randomized participants. Ongoing clinical benefit at Cycle 16 was summarized for overall participants, as due to switches in mode of administration up to Cycle 16, it would be impossible to isolate the effect of the randomization arms. Hence, per-arm data can't be presented.
Measure: Number; unit: percentage of participants
Groups:
- Atezolizumab: Participants received atezolizumab IV, 1200 mg and/or SC, 1875 mg Q3W up to Cycle 16 in Treatment Crossover Period and Treatment Continuation Period for participants with early-stage NSCLC or until loss of clinical benefit for participants with advanced NSCLC.
Arm/Group | Atezolizumab
Number analyzed (Participants) | 179
percentage of participants | 44.7

27. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is untoward medical occurrence in a participant administered a pharmaceutical product and regardless of causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with use of investigational product, whether or not considered related to the investigational product. Percentages have been rounded off.
Time Frame: Up to 90 days after the final dose of study drug (Up to 2.4 years)
Population: Safety evaluable population included all participants who received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Groups:
- Crossover Atezolizumab IV: Participants who were administered atezolizumab, IV infusion, 1200 mg, Q3W in Cycles 1 to 3 or Cycles 4 to 6 (cycle length=21 days), depending on the sequence (IV/SC or SC/IV) they were assigned in the Treatment Crossover Period are reported in this arm.
- Crossover Atezolizumab SC: Participants who were administered atezolizumab, SC injections, 1875 mg, Q3W for Cycles 1 to 3 or Cycles 4 to 6 (cycle length=21 days), depending on the sequence (IV/SC or SC/IV) they were assigned in the Treatment Crossover Period are reported in this arm.
- Continuation Atezolizumab IV: Participants in this arm chose to continue treatment with atezolizumab IV, 1200 mg Q3W up to Cycle 16 for participants with early-stage NSCLC or until loss of clinical benefit for participants with advanced NSCLC.
- Continuation Atezolizumab SC: Participants in this arm chose to continue treatment with atezolizumab SC, 1875 mg Q3W up to Cycle 16 for participants with early-stage NSCLC or until loss of clinical benefit for participants with advanced NSCLC.
Arm/Group | Crossover Atezolizumab IV | Crossover Atezolizumab SC | Continuation Atezolizumab IV | Continuation Atezolizumab SC
Number analyzed (Participants) | 160 | 155 | 26 | 89
percentage of participants | 59.4 | 47.7 | 76.9 | 67.4

28. Secondary Outcome: Percentage of Participants With AEs During Treatment Cross-over Period
Description: An AE is untoward medical occurrence in participant administered a pharmaceutical product and regardless of causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom/disease temporally associated with use of investigational product, whether or not considered related to investigational product. The safety of switching from atezolizumab SC to atezolizumab IV and from atezolizumab IV to atezolizumab SC is being assessed in this outcome measure. Percentages have been rounded off.
Time Frame: From Cycle 1 Day 1 up to Cycle 3 Day 21; From Cycle 4 Day 1 up to Cycle 6 Day 21 (cycle length=21 days)
Population: Safety evaluable population included all participants who received at least one dose of study treatment. In this analysis, participants were grouped by study arm and treatment period during the Crossover Period.
Measure: Number; unit: percentage of participants
Groups:
- Atezolizumab IV/ SC (Cycles 1 to 3): Participants were administered atezolizumab, IV infusion, 1200 mg, Q3W for Cycles 1 to 3 (cycle length=21 days) of the Treatment Crossover Period.
- Atezolizumab IV/SC (Cycles 4 to 6): Participants were administered atezolizumab, SC injections, 1875 mg, Q3W for Cycles 4 to 6 (cycle length=21 days) of the Treatment Crossover Period.
- Atezolizumab SC/IV (Cycles 1 to 3): Participants were administered atezolizumab, SC injections, 1875 mg, Q3W for Cycles 1 to 3 (cycle length=21 days) of the Treatment Crossover Period.
- Atezolizumab SC/IV (Cycles 4 to 6): Participants were administered atezolizumab, IV infusion, 1200 mg, Q3W for Cycles 4 to 6 (cycle length=21 days) of the Treatment Crossover Period.
Arm/Group | Atezolizumab IV/ SC (Cycles 1 to 3) | Atezolizumab IV/SC (Cycles 4 to 6) | Atezolizumab SC/IV (Cycles 1 to 3) | Atezolizumab SC/IV (Cycles 4 to 6)
Number analyzed (Participants) | 89 | 69 | 86 | 71
percentage of participants | 62.9 | 39.1 | 54.7 | 53.5

ADVERSE EVENTS:
Time Frame: Up to 90 days after the final dose of study drug (Up to 2.4 years)
Description: Safety evaluable population included all participants who received at least one dose of study treatment. As pre-planned, adverse events are presented for IV and SC administration of atezolizumab for each study period (crossover and continuation) and overall for all participants.
Groups:
- All Participants: This arm includes all participants who were administered atezolizumab IV, 1200 mg, and/or SC, 1875 mg Q3W up to Cycle 16 in the Treatment Crossover Period and Treatment Continuation Period for participants with early-stage NSCLC or until loss of clinical benefit for participants with advanced NSCLC.
Arm/Group | Crossover Atezolizumab IV | Crossover Atezolizumab SC | Continuation Atezolizumab IV | Continuation Atezolizumab SC | All Participants
All-Cause Mortality (participants affected / at risk) | 16/160 | 21/155 | 5/26 | 12/89 | 54/175
Serious Adverse Events (participants affected / at risk) | 15/160 | 13/155 | 6/26 | 12/89 | 45/175
Other Adverse Events (participants affected / at risk) | 60/160 | 52/155 | 16/26 | 44/89 | 172/175
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crossover Atezolizumab IV (N=160) | Crossover Atezolizumab SC (N=155) | Continuation Atezolizumab IV (N=26) | Continuation Atezolizumab SC (N=89) | All Participants (N=175)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Autoimmune myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated encephalitis (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 3 (4)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crossover Atezolizumab IV (N=160) | Crossover Atezolizumab SC (N=155) | Continuation Atezolizumab IV (N=26) | Continuation Atezolizumab SC (N=89) | All Participants (N=175)
Diarrhoea (Gastrointestinal disorders) | 9 (11) | 10 (10) | 4 (5) | 7 (10) | 24 (36)
Asthenia (General disorders) | 9 (9) | 8 (9) | 1 (1) | 6 (6) | 23 (25)
Injection site reaction (General disorders) | 0 (0) | 16 (24) | 0 (0) | 3 (3) | 19 (27)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (9) | 8 (8) | 0 (0) | 8 (13) | 21 (30)
Rash (Skin and subcutaneous tissue disorders) | 10 (10) | 4 (5) | 1 (1) | 5 (6) | 18 (22)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 3 (3) | 2 (2) | 1 (1) | 9 (9)
Hypothyroidism (Endocrine disorders) | 6 (6) | 1 (1) | 3 (3) | 3 (3) | 13 (13)
Fatigue (General disorders) | 6 (6) | 7 (7) | 2 (2) | 1 (1) | 14 (16)
Bronchitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 6 (6) | 9 (9)
COVID-19 (Infections and infestations) | 3 (3) | 2 (2) | 2 (2) | 4 (4) | 11 (11)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 2 (2) | 3 (4) | 7 (9)
Blood creatinine increased (Investigations) | 4 (5) | 4 (4) | 2 (2) | 6 (6) | 15 (17)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 2 (2) | 1 (1) | 10 (11)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (3) | 0 (0) | 7 (7) | 15 (18)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6) | 2 (2) | 3 (3) | 16 (16)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 1 (1) | 5 (5) | 9 (11)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7) | 2 (2) | 7 (7) | 21 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-02-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT05171777/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT05171777/SAP_001.pdf